CLINICAL TRIAL: NCT07382713
Title: Fluzoparib Combined With Famitinib as Maintenance Therapy After Response to First-Line Platinum-Based Chemotherapy in Patients With Advanced Ovarian Cancer: A Single-Arm, Multicenter Clinical Study
Brief Title: Fluzoparib Plus Famitinib Maintenance After First-Line Platinum Response in Advanced Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinhua Zhou (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jinhua Zhou, Director, Department of Obstetrics and Gynecology, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2026091
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib; famitinib

STUDY DESIGN:
Intervention Model Description: Single-group assignment: all participants receive fluzoparib + famitinib as post-first-line platinum response maintenance therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance Therapy: Fluzoparib + Famitinib (Experimental): Patients who achieved complete or partial response after first-line platinum-based chemotherapy receive maintenance therapy with fluzoparib plus famitinib malate. Fluzoparib is administered orally at 150 mg twice daily, and famitinib malate is administered orally at 10 mg once daily in 28-day cycles, continued until disease progression, unacceptable toxicity, withdrawal of consent, or completion of up to 24 cycles.
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib is administered orally at a dose of 150 mg twice daily, and famitinib malate is administered orally at a dose of 10 mg once daily. Treatment is given in 28-day cycles as maintenance therapy following complete or partial response to first-line platinum-based chemotherapy, and is continued until disease progression, unacceptable toxicity, withdrawal of consent, initiation of new anti-tumor therapy, or completion of up to 24 cycles.
  Other Names: Famitinib

SUMMARY:
This is a single-arm, open-label, multicenter exploratory clinical study designed to evaluate the efficacy and safety of fluzoparib combined with famitinib malate as maintenance therapy in patients with newly diagnosed advanced (FIGO III-IV) high-grade serous or endometrioid ovarian cancer (including fallopian tube and primary peritoneal cancer) who have achieved a complete response (CR) or partial response (PR) after first-line platinum-based chemotherapy (with or without bevacizumab). Eligible women aged 18-75 years with ECOG 0-1 will start study treatment within <9 weeks after the last platinum dose. Participants will receive fluzoparib 150 mg orally twice daily plus famitinib malate 10 mg orally once daily in 28-day cycles, continuing for up to 24 cycles or until disease progression, unacceptable toxicity, initiation of new anti-tumor therapy, withdrawal of consent, or investigator decision. The primary endpoint is progression-free survival (PFS); secondary endpoints include overall survival (OS), duration of response (DOR), time to response (TTR), and PFS-2.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18 to 75 years at the time of informed consent. Newly diagnosed, histologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer, including high-grade serous or high-grade endometrioid carcinoma.

FIGO stage III-IV disease at initial diagnosis. Achieved complete response (CR) or partial response (PR) after completion of first-line platinum-based chemotherapy, with or without bevacizumab.

Initiation of study treatment within 9 weeks after the last dose of platinum-based chemotherapy.

ECOG performance status 0-1. Adequate bone marrow, liver, and renal function, as defined by protocol-specified laboratory criteria.

Life expectancy of ≥12 weeks. Ability to swallow oral medications and comply with study requirements. Signed written informed consent prior to any study-specific procedures.

Exclusion Criteria:

Evidence of disease progression during or after first-line platinum-based chemotherapy.

Prior treatment with any PARP inhibitor or anti-angiogenic tyrosine kinase inhibitor (except bevacizumab as part of first-line therapy).

Prior systemic anti-cancer therapy for ovarian cancer other than first-line platinum-based chemotherapy.

Uncontrolled or significant cardiovascular disease, including but not limited to uncontrolled hypertension, recent myocardial infarction, or clinically significant arrhythmia.

Active or uncontrolled infection, or serious concomitant systemic disorders that may interfere with study participation.

Known central nervous system metastases. History of other malignancies within the past 5 years, except for adequately treated carcinoma in situ of the cervix or non-melanoma skin cancer.

Pregnant or breastfeeding women. Known hypersensitivity to fluzoparib, famitinib, or any of their excipients. Any condition that, in the investigator's judgment, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From treatment initiation up to approximately 48 months
  Progression-free survival is defined as the time from initiation of maintenance treatment with fluzoparib plus famitinib to the first documentation of disease progression according to RECIST v1.1 criteria or death from any cause, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data publicly available.